CLINICAL TRIAL: NCT01987427
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Pilot Study of 12-week Duration to Assess the Short-term Safety and Tolerability of Lorcaserin Plus Two Doses of Immediate-Release Phentermine-HCl Compared With Lorcaserin Alone in Overweight and Obese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-A001-402
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Chronic Weight Management
Keywords: Overweight; Obese; Weight Management
MeSH Terms: conditions — Overweight; Obesity | interventions — lorcaserin; Phentermine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): lorcaserin + phentermine placebo
  Interventions: Drug: lorcaserin + phentermine placebo
- B (Experimental): lorcaserin + phentermine-HCl + phentermine placebo
  Interventions: Drug: lorcaserin + phentermine-HCl + phentermine placebo
- C (Experimental): lorcaserin + phentermine-HCl
  Interventions: Drug: lorcaserin + phentermine-HCl

INTERVENTIONS:
Drug: lorcaserin + phentermine placebo — lorcaserin 10 mg BID + phentermine placebo BID
  Arms: A
Drug: lorcaserin + phentermine-HCl + phentermine placebo — lorcaserin 10 mg BID + phentermine-HCl 15 mg QD + phentermine placebo QD
  Arms: B
Drug: lorcaserin + phentermine-HCl — lorcaserin 10 mg BID + phentermine-HCl 15 mg BID
  Arms: C

SUMMARY:
APD356-A001-402 is a multicenter, double-blind, randomized, parallel-group pilot study of 12-week duration in overweight and obese adults. Approximately 225 subjects will be randomized to one of three treatment arms in a ratio 1:1:1 and will receive the combinations of lorcaserin 10 mg twice daily (BID) plus immediate-release phentermine-HCl 15 mg BID or 15 mg once daily (QD), or lorcaserin alone.

DETAILED DESCRIPTION:
All subjects will take lorcaserin and phentermine-HCl/placebo once in the morning and again in the mid-afternoon. The dosing is timed to help reduce potential insomnia due to phentermine. Subjects in Arm A will take one tablet twice daily of lorcaserin 10 mg in combination with one capsule twice daily of phentermine placebo. Subjects in Arm B will take one tablet twice daily of lorcaserin 10 mg, one capsule of phentermine-HCl 15 mg once daily in the morning, and one capsule of phentermine placebo once daily in the mid-afternoon. Subjects in Arm C will take one tablet twice daily of lorcaserin 10 mg in combination with one capsule twice daily of phentermine-HCl 15 mg. Subjects will be instructed to take lorcaserin tablets and phentermine/placebo capsules concurrently and attempt to remain on a consistent daily schedule. The study will recruit obese (body mass index [BMI] greater than or equal to 30 kg/m2) subjects with or without a weight-related comorbid condition (e.g., hypertension, dyslipidemia, or sleep apnea) or overweight (BMI greater than or equal to 27 to 29.9 kg/m2) subjects with at least one weight-related co-morbid condition. At least one third of the subjects will have a BMI of 40 kg/m2 or greater, because there is a high likelihood that this combination therapy will be used by these subjects in medical practice.

A lifestyle intervention program, using a 12-week adaptation of the Arena Healthy Lifestyles Program, including diet and exercise counseling, will be implemented for obesity/overweight.

Blood sampling will be performed to evaluate the pharmacokinetics (PK) of lorcaserin and phentermine using population PK modeling as well as the potential relationships between exposure to the lorcaserin/phentermine and measures of safety and change from baseline in body weight, using population PK/PD (pharmacodynamics) modeling.

ELIGIBILITY:
Inclusion Criteria

1. BMI is 30 kg/m2 or greater with or without a weight-related comorbid condition (e.g., hypertension, dyslipidemia, sleep apnea), or 27 to 29.9 kg/m2 with at least one weight-related comorbid condition.
2. Ambulatory and able to perform moderate exercise.
3. Male or female subjects between 18 and 60 years at the time of informed consent.
4. Provide written informed consent.
5. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria

1. Recent treatment (within 14 days of the Screening Visit and any time prior to randomization) with monoamine oxidase inhibitors (MAOIs). MAOIs have been associated with a risk of hypertensive crisis when used with phentermine.
2. Active or recent history (within 1 month prior to the Screening Visit) of major depression or other major psychiatric disease requiring treatment (i.e., within 1 month of the Screening Visit and any time prior to randomization or thereafter during the study) with prescription medication (e.g., SSRIs, SNRIs, tricyclics, antipsychotics, lithium, Wellbutrin).
3. Use of selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs) (including buproprion) for reasons other than active psychiatric indications (e.g., migraine, weight loss, smoking cessation) within 1 month prior to the Screening Visit).
4. Medication history that includes use of one or more of the following:

   1. Fenfluramine or related derivatives (i.e., dexfenfluramine, norfenfluramine)
   2. Agents that have documented correlation with increased incidence of valvulopathy and/or primary pulmonary hypertension (e.g., cabergoline, cyproheptadine, trazodone, nefazodone, amoxapine, mirtazapine, pergolide, ergotamine, methysergide)
5. Recent treatment (i.e., within 1 month of the Screening Visit and any time prior to randomization or thereafter during the study) with over-the-counter (OTC) weight loss products or appetite suppressants (including herbal weight loss agents), or within 6 months and any time prior to randomization or thereafter during the study, with a prescription weight loss drug (e.g., phentermine, phentermine/topiramate, orlistat).
6. Use of St. John's Wort within 1 month prior to the Screening Visit and for the duration of the study. St. John's Wort has been associated with serotonin syndrome when used with another serotonergic drug.
7. Hypersensitivity to sympathomimetic amines or the study drugs.
8. History of stroke, transient ischemic attack, arrhythmias, congestive heart failure, and/or peripheral vascular disease.
9. Recent history of active cardiovascular disease, including chronic stable angina or an unstable angina episode or myocardial infarction within the 3 months prior to the Screening Visit.
10. Uncontrolled hypertension defined as systolic blood pressure greater than or equal to 150 or diastolic blood pressure greater than or equal to 95 on 2 readings taken on different days. Subjects who have uncontrolled hypertension at screening may be re-screened greater than 1 month following initiation or adjustment of antihypertensive therapy.
11. History of or active pulmonary artery hypertension.
12. Severe renal impairment (creatinine clearance less than 30 mL/min, as calculated by the Cockroft-Gault equation based on ideal body weight) or end stage renal disease.
13. History of valve replacement surgery; clinically significant valvular stenosis; history of or active clinically significant valvulopathy (defined as aortic insufficiency of mild, moderate, or severe intensity and/or mitral insufficiency of moderate or severe intensity).
14. History of or active (confirmed fasting glucose greater than 126 mg/dL or hemoglobin A1c [HbA1c] greater than ULN [6.5% at central laboratory]) diabetes mellitus (type I, II or other) and/or currently taking medications for type I or II diabetes. A past history of gestational diabetes that has resolved is permissible.
15. Glaucoma.
16. Abnormal thyroid stimulating hormone (TSH) laboratory value greater than 1.5 x Upper Limit of Normal (ULN)
17. Hyperthyroidism, including abnormal screening laboratory values with T3 greater than ULN and TSH less than Lower Limit of Normal (LLN), and subjects taking methimazole or propylthiouracil (PTU) and/or beta-blockers for hyperthyroidism.
18. Recent history (within 2 years prior to the Screening Visit) of alcohol or drug/solvent abuse or a positive screen for drugs of abuse at screening.
19. Significant change is smoking habits or tobacco product use within 3 months prior to the Screening Visit.
20. Use of tobacco products (i.e., smokes more than one-half pack of cigarettes per day, or smokes more than 2 cigars per day, or uses 3 or more pinches of smokeless tobacco per day).
21. Surgical procedure for the treatment of obesity (i.e., gastric bypass, gastric banding), even if reversed prior to screening.
22. Planned surgery during the study period that may interfere with completion or compliance with the protocol.
23. A prolonged QT/QTc interval (QTc Bazett's greater than 450 msec) as demonstrated by a repeated electrocardiogram (ECG).
24. Participation in any clinical study with an investigational drug, biologic, or device within 1 month prior to screening.
25. Significant change in diet or level of physical activity within 1 month prior to dosing that in the opinion of the investigator(s) may confound the results of the study.
26. Change in weight of greater than 5 kg within 3 months of screening.
27. Use of a very-low calorie (less than 800/day) liquid weight loss diet within 6 months prior to screening and any time prior to randomization.
28. Eligible male and female subjects participating in a conception process (i.e., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
29. Females who are lactating or pregnant at Screening or Baseline Visit (as documented by a negative serum or urine pregnancy test with a minimum sensitivity of 25 IU/L or equivalent units of beta-human chorionic gonadotropin [B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
30. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least one month before dosing).
31. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation. Females not meeting these criteria will be excluded from the study.
32. Any medical or other condition that in the opinion of the investigator(s) would preclude the subject's participation in a clinical study, such as significantly abnormal laboratory results or any physical or mental condition that prevents compliance with the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Radiant Research - Arizona, Chandler, Arizona
  - Scripps Clinical Research Center, La Jolla, California
  - Translational Research Institute for Metabolism and Diabetes, Orlando, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Weill Cornell College, New York, New York
  - Duke University, Durham, North Carolina
  - Radiant Research - Columbus, Columbus, Ohio
  - Radiant Research - South Carolina, Anderson, South Carolina
  - Radiant Research - Dallas, Dallas, Texas
  - National Clinical Research - Norfolk, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Rebello CJ, Nikonova EV, Zhou S, Aronne LJ, Fujioka K, Garvey WT, Smith SR, Coulter AA, Greenway FL. Effect of Lorcaserin Alone and in Combination with Phentermine on Food Cravings After 12-Week Treatment: A Randomized Substudy. Obesity (Silver Spring). 2018 Feb;26(2):332-339. doi: 10.1002/oby.22094. PMID 29363287
- [Derived] Smith SR, Garvey WT, Greenway FL, Zhou S, Fain R, Pilson R, Fujioka K, Aronne LJ. Coadministration of lorcaserin and phentermine for weight management: A 12-week, randomized, pilot safety study. Obesity (Silver Spring). 2017 May;25(5):857-865. doi: 10.1002/oby.21811. PMID 28440045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 sites in the United States from 30 October 2013 to 03 September 2014.
Pre-assignment Details: A total of 344 participants were screened and enrolled, of which 106 were screen failures and 238 were randomized to receive study treatment, out of which 235 participants were treated.
Groups:
- Lorcaserin 10 mg BID + Phentermine Placebo BID: Participants received lorcaserin 10 milligram (mg) tablet along with phentermine placebo-matching capsule, orally, twice daily (BID) for 12 weeks.
- Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD: Participants received lorcaserin 10 mg tablet, orally, BID along with phentermine 15 mg capsule, orally, once daily (QD), and phentermine placebo-matching capsule, orally, QD for 12 weeks.
- Lorcaserin 10 mg BID + Phentermine 15 mg BID: Participants received lorcaserin 10 mg tablet along with phentermine 15 mg capsule, orally, BID for 12 weeks.
Period: Overall Study
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Started | 78 | 78 | 79
Completed | 64 | 68 | 59
Not Completed | 14 | 10 | 20
Not completed — Adverse Event | 4 | 2 | 8
Not completed — Lost to Follow-up | 6 | 6 | 9
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least one dose of the study drug.
Groups:
- Lorcaserin 10 mg BID + Phentermine Placebo BID: Participants received lorcaserin 10 mg tablet along with phentermine placebo-matching capsule, orally, BID for 12 weeks.
- Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD: Participants received lorcaserin 10 mg tablet, orally, BID along with phentermine 15 mg capsule, orally, QD, and phentermine placebo-matching capsule, orally, QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID | Total
Number analyzed (Participants) | 78 | 78 | 79 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.02) | 44.8 (11.08) | 41.2 (11.69) | 42.8 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 70 | 62 | 200
  Male | 10 | 8 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 6 | 24
  Not Hispanic or Latino | 67 | 71 | 73 | 211
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 29 | 26 | 32 | 87
  White | 46 | 50 | 44 | 140
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting at Least One of Nine Adverse Events (AEs) of Main Interests That May Related to Serotonergic Reaction
Description: The nine common serotonergic AEs were headache, dizziness, nausea, fatigue, dry mouth, diarrhea, vomiting, insomnia, and/or anxiety.
Time Frame: Baseline up to Week 12 (end of treatment)
Population: The full analysis set included all randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
percentage of participants | 37.2 | 42.3 | 40.5

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and AEs Leading to Study Drug Discontinuation
Time Frame: Baseline up to Week 16
Population: The safety analysis set included all randomized participants who received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
Participants
  TEAE | 50 | 52 | 54
  SAE | 0 | 2 | 1
  AEs leading to study drug discontinuation | 4 | 2 | 9

3. Secondary Outcome: Number of Participants With Treatment-Emergent Markedly Abnormal Laboratory Values
Time Frame: Baseline up to Week 16
Population: The safety analysis set included all randomized participants who received at least one dose of study drug and had at least one post-baseline safety assessment. Participants who were evaluable for this measure for given laboratory parameter were included in the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
Participants
  Gamma glutamyl transferase: high: number analyzed (Participants) | 72 | 76 | 73
  Gamma glutamyl transferase: high | 0 | 1 | 1
  Phosphorus: low: number analyzed (Participants) | 72 | 76 | 73
  Phosphorus: low | 0 | 1 | 0
  Potassium: high: number analyzed (Participants) | 72 | 76 | 73
  Potassium: high | 1 | 3 | 1
  Total bilirubin: high: number analyzed (Participants) | 72 | 76 | 73
  Total bilirubin: high | 0 | 1 | 0
  Triglycerides: High: number analyzed (Participants) | 72 | 76 | 73
  Triglycerides: High | 0 | 1 | 0
  Uric acid: high: number analyzed (Participants) | 72 | 76 | 73
  Uric acid: high | 1 | 0 | 0
  Hemoglobin: low: number analyzed (Participants) | 72 | 77 | 73
  Hemoglobin: low | 1 | 1 | 0
  Lymphocytes: high: number analyzed (Participants) | 72 | 77 | 73
  Lymphocytes: high | 0 | 0 | 1
  Neutrophils: low: number analyzed (Participants) | 72 | 77 | 73
  Neutrophils: low | 2 | 1 | 0
  White blood cell (WBC) count: low: number analyzed (Participants) | 72 | 77 | 73
  White blood cell (WBC) count: low | 0 | 0 | 1

4. Secondary Outcome: Mean Change From Baseline in Body Weight at Weeks 1, 2, 4, 8, and 12
Time Frame: Baseline, Weeks 1, 2, 4, 8 and 12
Population: The Modified Intent-to-Treat (MITT) set included all randomized participants who received at least one dose of the study drug and had a Baseline weight measurement and a post-randomization weight measurement. Participants who were evaluable for this measure at given time period were included in the assessment.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
kilogram (kg)
  Baseline | 105.33 (20.994) | 105.04 (23.399) | 106.63 (19.703)
  Change at Week 1: number analyzed (Participants) | 75 | 74 | 79
  Change at Week 1 | -0.94 (1.290) | -1.36 (1.341) | -1.97 (1.477)
  Change at Week 2: number analyzed (Participants) | 78 | 77 | 79
  Change at Week 2 | -1.56 (1.547) | -2.43 (1.566) | -2.94 (1.925)
  Change at Week 4 | -2.27 (1.823) | -3.81 (2.442) | -4.44 (2.606)
  Change at Week 8 | -2.87 (2.691) | -5.76 (3.711) | -6.33 (3.913)
  Change at Week 12 | -3.48 (3.727) | -7.00 (5.950) | -7.55 (4.725)

5. Secondary Outcome: Percent Change From Baseline in Body Weight at Weeks 1, 2, 4, 8, and 12
Time Frame: Baseline, Weeks 1, 2, 4, 8 and 12
Population: The MITT set included all randomized participants who received at least one dose of the study drug and had a Baseline weight measurement and a post-randomization weight measurement. Participants who were evaluable for this measure at given time period were included in the assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
percent change
  Week 1: number analyzed (Participants) | 75 | 74 | 79
  Week 1 | -0.93 (1.212) | -1.28 (1.234) | -1.82 (1.358)
  Week 2: number analyzed (Participants) | 78 | 77 | 79
  Week 2 | -1.47 (1.451) | -2.33 (1.465) | -2.75 (1.787)
  Week 4 | -2.18 (1.744) | -3.68 (2.265) | -4.20 (2.459)
  Week 8 | -2.77 (2.551) | -5.54 (3.466) | -6.03 (3.722)
  Week 12 | -3.29 (3.363) | -6.69 (5.377) | -7.23 (4.611)

6. Secondary Outcome: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 5 Percent (%) Weight Reduction at Week 12
Time Frame: Week 12 (end of treatment)
Population: The MITT set included all randomized participants who received at least one dose of the study drug and had a Baseline weight measurement and a post-randomization weight measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
percentage of participants | 28.2 | 59.0 | 70.9

7. Secondary Outcome: Change From Baseline in Waist Circumference and Hip Circumference at Week 12
Time Frame: Baseline and Week 12 (end of treatment)
Population: The MITT population consisted of all randomized participants who received at least one dose of the study drug and had a Baseline weight measurement and a post-randomization weight measurement. Participants who were evaluable for this measure at given time period were included in the assessment.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
centimeter (cm)
  Waist Circumference: Baseline | 112.2 (13.82) | 112.2 (15.09) | 114.0 (12.02)
  Waist Circumference: Change at Week 12: number analyzed (Participants) | 57 | 66 | 57
  Waist Circumference: Change at Week 12 | -3.4 (7.98) | -4.7 (10.31) | -7.1 (5.53)
  Hip Circumference: Baseline | 124.1 (14.30) | 123.7 (14.27) | 125.4 (12.81)
  Hip Circumference: Change at Week 12: number analyzed (Participants) | 57 | 66 | 57
  Hip Circumference: Change at Week 12 | -2.8 (8.05) | -3.6 (11.29) | -6.2 (4.41)

8. Secondary Outcome: Change From Baseline in Waist to Hip Circumference Ratio at Week 12
Time Frame: Baseline and Week 12 (end of treatment)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
Number analyzed (Participants) | 78 | 78 | 79
ratio
  Baseline | 0.91 (0.083) | 0.91 (0.091) | 0.91 (0.084)
  Change at Week 12: number analyzed (Participants) | 57 | 66 | 57
  Change at Week 12 | -0.01 (0.102) | -0.01 (0.044) | -0.01 (0.036)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Baseline) up to Week 16 (30 days after last dose of study drug on Week 12/end of treatment)
Arm/Group | Lorcaserin 10 mg BID + Phentermine Placebo BID | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD | Lorcaserin 10 mg BID + Phentermine 15 mg BID
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 2/78 | 1/79
Other Adverse Events (participants affected / at risk) | 50/78 | 51/78 | 54/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin 10 mg BID + Phentermine Placebo BID (N=78) | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD (N=78) | Lorcaserin 10 mg BID + Phentermine 15 mg BID (N=79)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin 10 mg BID + Phentermine Placebo BID (N=78) | Lorcaserin 10mg BID+Phentermine 15mg QD+Phentermine Placebo QD (N=78) | Lorcaserin 10 mg BID + Phentermine 15 mg BID (N=79)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 7 | 11
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 21 | 18
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 6
Salivary gland pain (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 3
Chest discomfort (General disorders) | 0 | 0 | 1
Chills (General disorders) | 2 | 1 | 0
Energy increased (General disorders) | 0 | 0 | 1
Eye complication associated with device (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 8 | 3 | 5
Feeling cold (General disorders) | 0 | 0 | 1
Feeling jittery (General disorders) | 1 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 2 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Perfume sensitivity (Immune system disorders) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Periorbital contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 8
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 14 | 7 | 11
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 2
Nerve root compression (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Bruxism (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 4 | 2
Loss of libido (Psychiatric disorders) | 0 | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No